CLINICAL TRIAL: NCT06032637
Title: Difference Between Pfannenstiel Incision and Higher Transverse Supra Umbilical Incision, During Elective Cesarean Section in Morbidly Obese Patients
Brief Title: Best Incision in Cesarean Section of Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, lecturer and consultant at Obstetrics and Gynecology Department., Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Obstet1222
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Morbid Obesity; Cesarean Section Complications
Keywords: elective cesarean section; morbid obesity; Pfannenstiel incision; Transverse supra-umbilical incision
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pfannenstiel incision (Active Comparator): Patients randomized to the Pfannenstiel incision arm will undergo a transverse skin incision 2-3cm above the symphysis pubis. Subcutaneous tissue will be dissected until anterior rectus sheath is exposed. A transverse incision will be made through the rectus sheath in line with the skin incision, avoiding injury to the inferior epigastric arteries. Rectus muscles will be separated manually along midline using blunt dissection. The peritoneum will be incised transversely and the hysterotomy extended laterally with uterine traction to deliver fetus. The visceral peritoneum will not be closed. Rectus muscles will not be re-approximated. Subcutaneous tissue will not be irrigated. Subcutaneous tissue will be closed if over 2cm depth. Skin will be closed with non-absorbable suture subcuticularly.
  Interventions: Procedure: Pfannenstiel incision
- Supra-Umbilical (Experimental): Patients randomized to the supra-umbilical transverse incision arm will undergo a transverse skin incision halfway between the umbilicus and xiphoid process, extending laterally to the semilunar lines. Subcutaneous tissue will be bluntly dissected until anterior rectus sheath is exposed. A transverse incision will be made through the rectus sheath in line with the skin incision, avoiding injury to the superior epigastric vessels. Rectus muscles will be split manually along midline using blunt dissection. The peritoneum will be incised transversely and the hysterotomy extended laterally with uterine traction to deliver fetus. The visceral peritoneum will not be closed. Rectus muscles will not be re-approximated. Subcutaneous tissue will not be irrigated. Subcutaneous tissue will be closed if over 2cm depth. Skin will be closed with non-absorbable suture subcuticularly.
  Interventions: Procedure: Supra-umbilical transverse incision

INTERVENTIONS:
Procedure: Pfannenstiel incision — Patients randomized to the supra-umbilical transverse incision arm will receive a transverse skin incision halfway between the umbilicus and xiphoid process, extending laterally to the semilunar lines. The subcutaneous tissue will be bluntly dissected until the anterior rectus sheath is exposed. A transverse incision will be made through the rectus sheath in line with the skin incision, avoiding injury to the superior epigastric vessels. The rectus muscles will be split manually using blunt dissection. The peritoneum will be incised transversely and the hysterotomy extended laterally to deliver the fetus. The visceral peritoneum will not be closed. The rectus muscles will not be re-approximated. The subcutaneous tissue will not be irrigated but closed if over 2cm depth. The skin will be closed with non-absorbable suture subcuticularly.
  Arms: Pfannenstiel incision
Procedure: Supra-umbilical transverse incision — Patients randomized to the supra-umbilical transverse incision arm will receive a transverse skin incision 3-4cm above the umbilicus, extending laterally to the semilunar lines, without panniculus retraction. The subcutaneous tissue will be bluntly dissected until the anterior rectus sheath is exposed. The rectus sheath will be incised transversely using electrocautery for hemostasis, avoiding injury to the superior epigastric vessels. The rectus muscles will be split manually along the midline using blunt dissection. The peritoneum will be transversely incised and the hysterotomy extended laterally to deliver the fetus. The visceral peritoneum will not be closed. The rectus muscles will not be re-approximated. The subcutaneous tissue will not be irrigated but closed if over 2cm depth. The skin will be closed with non-absorbable suture subcuticularly.
  Arms: Supra-Umbilical

SUMMARY:
The goal of this comparative clinical trial is to compare Pfannenstiel incision and higher transverse supra umbilical incision techniques during elective cesarean section in morbidly obese patients. The main questions it aims to answer are:

Is there a difference in operative time between the two incision techniques? Is there a difference in estimated blood loss between the two techniques? Is there a difference in post-operative pain scores between the two techniques? Is there a difference in wound complication rates between the two techniques? Participants will be randomly assigned to receive either a Pfannenstiel incision or a higher transverse supra umbilical incision during their scheduled cesarean delivery.

Researchers will compare the Pfannenstiel incision group to the higher transverse supra umbilical incision group to see if there are differences in operative time, blood loss, post-operative pain, and wound complications.

DETAILED DESCRIPTION:
This randomized controlled trial will enroll 60 morbidly obese pregnant patients scheduled for elective cesarean delivery at gestational age ≥37 weeks. Morbid obesity will be defined as pre-pregnancy body mass index ≥40 kg/m2.

Patients will be randomly allocated to one of two groups (30 patients per group):

Group 1 (Pfannenstiel group): Patients will undergo a transverse infraumbilical skin incision 2-3 cm above the symphysis pubis, followed by transverse incision of the anterior rectus sheath in the same line as the skin incision, blunt digital separation of the rectus muscles, and transverse uterine incision in the lower segment.

Group 2 (Supra-umbilical transverse group): Patients will undergo a transverse skin incision halfway between the umbilicus and xiphoid process, followed by transverse incision of the anterior rectus sheath in the same line, blunt digital separation of the rectus muscles, and transverse uterine incision in the lower segment.

The primary outcome measures will be operative time, estimated blood loss, post-operative pain scores, and wound complication rates. Secondary outcomes will include length of hospital stay, patient satisfaction scores, and cosmetic results.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 20 and 40 years.
* Singleton pregnancy.
* Gestational age ≥ 37 weeks.
* Scheduled for elective cesarean delivery.
* Morbid obesity, defined as pre-pregnancy body mass index (BMI) ≥ 40 kg/m2.
* Willing and able to provide informed consent.
* Able to adhere to study procedures and follow-up schedule.

Exclusion Criteria:

* Emergency cesarean delivery.
* Multiple gestation (twins, triplets, etc)
* Placenta previa or vasa previa.
* History of more than 1 previous cesarean delivery.
* HIV, hepatitis B/C infection.
* Current anticoagulation therapy.
* Immune-compromised conditions.
* Premature rupture of membranes.
* Pre-existing skin conditions affecting the abdomen.
* Inability to provide informed consent.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study will enroll only female participants, as the surgical procedures being compared are specific to cesarean delivery. Only pregnant patients who are scheduled to undergo elective cesarean section will be included. This study is restricted to women only given the gender-specific nature of pregnancy and childbirth. Patients must be female sex at birth with intact uteri in order to be eligible. Transgender male patients and individuals with no female reproductive organs will be excluded. Enrollment is limited to cisgender women only.
Enrollment: 60 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Rate of surgical site wound infection | 4 weeks after the surgery.
  Surgical site infections will be assessed at the cesarean incision site and tracked for 4 weeks postoperatively. Wound infection will be defined as purulent drainage from the incision, positive culture, and/or at least two of the following signs or symptoms: pain or tenderness, localized swelling, redness, or heat. The 4-week timeframe starts on the day of surgery (day 0) and ends 28 days postoperatively. Wound infections occurring up to 4 weeks after surgery will be captured and recorded as the primary outcome measure. Wound assessments will be performed daily during the hospital stay, at the post-op visit around 2 weeks, and at the 4-week follow-up visit.

SECONDARY OUTCOMES:
Operative time | during the surgery
  Operative time will be defined as the time from skin incision to complete wound closure. It will be recorded in minutes by a study investigator observing each procedure.
Hospital length of stay | From day of surgery to discharge, up to 8 weeks.
  Hospital length of stay will be defined as the number of days from surgery until discharge from the hospital.
Estimated blood loss | during the procedure
  Estimated blood loss will be assessed by the anesthesiologist and surgeon at the end of the procedure, based on the amount of blood in the suction canister and blood-soaked sponges/lap pads.
Postoperative pain | From end of surgery through 4 weeks postoperatively
  Postoperative pain will be assessed using a visual analog scale (VAS) of 0-10, with 0 being no pain and 10 being worst possible pain. Patients will rate their pain level at set intervals after surgery - immediately after recovery room discharge, daily while inpatient, and at 2 weeks and 4 weeks postop during follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Muhamed A Alhagrasy, M.D., Principal Investigator — Al-Azhar University
Locations (1):
- Al-Hussein University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The study involves a vulnerable population of pregnant women and collecting sensitive health information. Sharing individual participant data could risk participant privacy and confidentiality even if de-identified.
  The sample size is small at only 60 participants. individual participant data from such a small sample has a higher risk of re-identification.
  The research team intends to use the individual participant data for additional analyses and future studies. Sharing individual participant data may lead to misuse, misinterpretation, or compromised validity if not properly analyzed.
  Logistical barriers make preparing and curating a database for individual participant data sharing highly resource and time intensive for the research team.